CLINICAL TRIAL: NCT02379416
Title: Phase I Trial of the Combination of Nilotinib and Paclitaxel in Adults and Pediatric Patients With Refractory Solid Tumors
Brief Title: Combination Nilotinib and Paclitaxel in Adults With Relapsed Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 150086; 15-C-0086
Record Dates: First submitted 2015-03-04; First posted 2015-03-05 (Estimated); Last update posted 2025-08-26 (Actual); Status verified 2025-08-21

CONDITIONS: Solid Tumors
Keywords: Drug Efflux; Taxanes; Combination; Bcr-Abl Kinase Inhibitors; Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — nilotinib; Paclitaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment (Experimental): The starting dose of nilotinib will be administered at 300 mg orally BID from cycle 1 day 2 and paclitaxel will be administered IV at 60 mg/m2 at dose level 1 on Days 1, 8, and 15 in 28-day cycles. For cycle 2 on, nilotinib will be administered from day 1. Dose escalation will follow a 3+3 design, with dose limiting toxicities defined during cycle 1.
  Interventions: Drug: Nilotinib + Paclitaxel

INTERVENTIONS:
Drug: Nilotinib + Paclitaxel — The BCR-Abl kinase inhibitor nilotinib demonstrated greater than additive activity in combination with the anti-tubulin agent paclitaxel in preclinical xenograft models, justifying the clinical evaluation of this combination for its antitumor activity

SUMMARY:
Background:

- Researchers want to find better ways to treat cancer. One drug that treats cancer is paclitaxel. Sometimes proteins block that drug from working. Researchers want to see if another drug, nilotinib, helps paclitaxel work better.

Objective:

- To test the safety of nilotinib plus paclitaxel and find out what doses of the drugs can be given safely to people.

Eligibility:

- Adults at least 18 years old with advanced cancer that has progressed after receiving standard treatment, or for which no effective therapy exists.

Design:

* Participants will be screened with tests they usually get in their cancer care: medical history, physical exam, blood and urine tests, heart test, and scans.
* Participants will take the two study drugs in 28-day cycles. They will keep a medicine diary.
* Nilotinib will be taken by mouth twice every day except day 1 of the first cycle.
* Paclitaxel will be given by IV once a week for the first 3 weeks of a cycle. This will usually be done at the clinic.
* Most participants will have a weekly study visit every week for cycle 1, then the first 3 weeks of other cycles. They will have:
* Physical exam at every visit.
* Blood tests multiple times for cycle 1, then the first 3 weeks of other cycles.
* Scans every 8 weeks. These may be CT or MRI scans, in a machine that takes pictures. Or they may be ultrasounds, where a wand is pressed on the skin with gel on it.
* Around 30 days after stopping the study drugs, participants will be called to discuss any side effects.

DETAILED DESCRIPTION:
Background:

-The BCR-Abl kinase inhibitor nilotinib demonstrated greater than additive activity in combination with the anti-tubulin agent paclitaxel in preclinical xenograft models, justifying the clinical evaluation of this combination for its antitumor activity

Objectives:

* To establish the safety, tolerability, and maximum tolerated dose (MTD) of nilotinib plus paclitaxel in patients with refractory solid tumors, both in adult subjects >=18 years of age and in pediatric/adolescent subjects 12-17 years of age
* To determine the pharmacokinetics of paclitaxel and nilotinib when administered in combination
* To evaluate the pharmacodynamic effects of the combination on biomarkers of apoptosis, DNA damage response, and epithelial-to-mesenchymal transition

Eligibility:

* Study participants must have histologically confirmed solid tumor that has progressed on standard therapy known to prolong survival or for which no standard treatment options exist
* Age greater than or equal to 12
* No major surgery, radiation, or chemotherapy within 3 weeks prior to entering the study (6 weeks for nitrosoureas and mitomycin C).
* Adequate organ function

Study Design:

* This is an open-label Phase I trial
* During dose escalation, the starting dose of nilotinib will be administered at 300 mg orally BID from cycle 1 day 2 and paclitaxel will be administered IV at 60 mg/m2 at dose level 1 on Days 1, 8, and 15 in 28-day cycles. For cycle 2 on, nilotinib will be administered from day 1. Dose escalation will follow a 3+3 design, with dose limiting toxicities defined during cycle 1.
* Up to 33 adult patients will be accrued to a PD expansion phase at the MTD to further assess pharmacodynamic endpoints in tumor and CTCs.
* As of Amendment O (May 2020), patients ages 12-17 will be accrued to a separate pediatric expansion cohort to evaluate the safety, pharmacokinetics, and pharmacodynamics of this combination for pediatric patients.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patients must have histologically confirmed solid tumors that have progressed on standard therapy known to prolong survival or for which no standard treatment options exist.
* Age greater than or equal to 12 years.
* ECOG performance status less than or equal to 2.
* Life expectancy of greater than 3 months
* Patients must have normal organ and marrow function as defined below:

  * Absolute neutrophil count greater than or equal to 1,500/mcL
  * Platelets greater than or equal to 100,000/mcL
  * Total bilirubin less than or equal to 1.5 X institutional ULN (with the exception of those with Gilbert syndrome, who must have total bilirubin <=3 X institutional ULN)
  * AST(SGOT)/ALT(SGPT) less than or equal to 3 X institutional upper limit of normal; 5.0 x ULN in patients with liver metastases
  * creatinine less than or equal to 1.5 X institutional ULN OR
  * creatinine clearance greater than or equal to 60 mL/min/1.73 m2 for patients with creatinine levels greater than 1.5 mg/dL
* Nilotinib and paclitaxel have both been assigned to pregnancy category D by the FDA. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation and for at least 3 months after dosing with study drugs ceases. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 3 months after completion of study drug administration.
* Patients must have completed radiation therapy, or major surgery greater than or equal to 3 weeks, or biologic therapy or chemotherapy greater than or equal to 5 half-lives or 3 weeks, whichever is shorter (6 weeks for nitrosoureas and mitomycin C) prior to entering the study. Patients must be greater than or equal to 2 weeks since any prior administration of a study drug in a Phase 0 or equivalent study and be greater than or equal to1 week from palliative radiation therapy. Patients must have recovered to eligibility levels from prior toxicity or adverse events. Treatment with bisphosphonates is permitted.
* For the PD-expansion cohort, patients must be willing to give biopsies for research and have tumors amenable for the acceptable biopsy procedures- or in lieu of baseline biopsies, patient must have and be willing to submit at registration archival tumor biopsy tissue from a previous research study or medical care. Criteria for the submission of archival tissue are:
* Tissue must have been collected within 3 months prior to registration.
* Patient must not have received any intervening therapy for their cancer since the collection of the tumor sample.
* Tumor tissue must meet the minimum requirements

EXCLUSION CRITERIA:

* QTcF interval of less than 450 msec at study entry; congenital long QT syndrome
* Sensory/motor neuropathy less than or equal to Grade 2
* Patients who are receiving any other investigational agents.
* Patients with active brain metastases or carcinomatous meningitis are excluded from this clinical trial. Patients with treated brain metastases, whose brain metastatic disease has remained stable for less than or equal to 4 weeks without requiring steroid and anti-seizure medication are eligible to participate.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to study drugs.
* Uncontrolled intercurrent illness including, but not limited to, serious untreated infection, symptomatic respiratory failure/congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because nilotinib and paclitaxel have been assigned to pregnancy category D by the FDA. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with the study drugs, breastfeeding should be discontinued prior to the first dose of study drug and women should refrain from nursing throughout the treatment period and for 3 months following the last dose of study drug.
* HIV-positive patients on combination antiretroviral therapy are ineligible because of possible PK interactions with study drugs.
* Both men and women of all races and ethnic groups are eligible for this trial.

Ages: 12 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2015-04-13 (Actual); Primary Completion 2026-06-27 (Estimated); Study Completion 2026-06-27 (Estimated)

PRIMARY OUTCOMES:
To establish the safety, tolerability, and maximum tolerated dose (MTD) of nilotinib plus paclitaxel combination in patients with refractory solid tumors | Cycle 1
  Safety, tolerability, and maximum tolerated dose (MTD) of nilotinib plus paclitaxel combination in patients with refractory solid tumors

SECONDARY OUTCOMES:
To determine the pharmacokinetics of paclitaxel when administered in combination with nilotinib | Cycle 1

CONTACTS AND LOCATIONS:
Overall Officials: Alice P Chen, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Kummar S, Chen HX, Wright J, Holbeck S, Millin MD, Tomaszewski J, Zweibel J, Collins J, Doroshow JH. Utilizing targeted cancer therapeutic agents in combination: novel approaches and urgent requirements. Nat Rev Drug Discov. 2010 Nov;9(11):843-56. doi: 10.1038/nrd3216. Epub 2010 Oct 29. PMID 21031001
- [Background] Tiwari AK, Sodani K, Dai CL, Abuznait AH, Singh S, Xiao ZJ, Patel A, Talele TT, Fu L, Kaddoumi A, Gallo JM, Chen ZS. Nilotinib potentiates anticancer drug sensitivity in murine ABCB1-, ABCG2-, and ABCC10-multidrug resistance xenograft models. Cancer Lett. 2013 Jan 28;328(2):307-17. doi: 10.1016/j.canlet.2012.10.001. Epub 2012 Oct 9. PMID 23063650
- [Background] Shen T, Kuang YH, Ashby CR, Lei Y, Chen A, Zhou Y, Chen X, Tiwari AK, Hopper-Borge E, Ouyang J, Chen ZS. Imatinib and nilotinib reverse multidrug resistance in cancer cells by inhibiting the efflux activity of the MRP7 (ABCC10). PLoS One. 2009 Oct 20;4(10):e7520. doi: 10.1371/journal.pone.0007520. PMID 19841739
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2015-C-0086.html